CLINICAL TRIAL: NCT00744094
Title: The Influence of Resistance Training on Body Composition and Muscle Characteristics in Healthy Elderly
Brief Title: Resistance Training in Elderly
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: The Anna Foundation (Other); DSM Food Specialties (Industry)
Responsible Party: Dr. L. van Loon, Maastricht University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MEC 06-3-062B
Record Dates: First submitted 2008-08-28; First posted 2008-08-29 (Estimated); Last update posted 2015-09-23 (Estimated); Status verified 2008-08

CONDITIONS: Sarcopenia; Atrophy; Aging
Keywords: resistance training; protein supplementation; hypertrophy
MeSH Terms: conditions — Sarcopenia; Atrophy; Hypertrophy | interventions — Resistance Training

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Placebo Comparator): placebo drink
  Interventions: Behavioral: Resistance training
- 2 (Experimental): protein drink
  Interventions: Dietary Supplement: protein drink; Behavioral: Resistance training

INTERVENTIONS:
Dietary Supplement: protein drink — 250 ml protein hydrolysate solution
  Arms: 2
Behavioral: Resistance training — 12 weeks resistance training, 3 days per week

SUMMARY:
In the present study the investigators aim to determine whether protein supplementation can augment the response to a 12 week resistance training program in healthy elderly men.

ELIGIBILITY:
Inclusion Criteria:

* Living independently

Exclusion Criteria:

* Diabetes
* Cardiovascular disease
* Orthopedic limitations
* Any disorder known to compromise ability for resistance training
* History of resistance training in past 5 years

Ages: 65 Years to 85 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 26 (Actual)
Dates: Start 2007-01; Primary Completion 2007-09 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Muscle mass measured at limb and cellular level | before and after 12 weeks of intervention

SECONDARY OUTCOMES:
Muscle strength | before and after 12 weeks of intervention
Body composition | before and after 12 weeks of intervention

CONTACTS AND LOCATIONS:
Overall Officials: Luc JC van Loon, PhD, Principal Investigator — Maastricht University
Locations (1):
- Maastricht University, Maastricht, Netherlands

REFERENCES:
- [Derived] Verdijk LB, Jonkers RA, Gleeson BG, Beelen M, Meijer K, Savelberg HH, Wodzig WK, Dendale P, van Loon LJ. Protein supplementation before and after exercise does not further augment skeletal muscle hypertrophy after resistance training in elderly men. Am J Clin Nutr. 2009 Feb;89(2):608-16. doi: 10.3945/ajcn.2008.26626. Epub 2008 Dec 23. PMID 19106243